CLINICAL TRIAL: NCT02446171
Title: An Open-Label, Randomized, 4-Period, 4-Treatment, Crossover, Single-Center, Single-Dose Bioavailability Study With Alternate Methods of Administration of Crushed Naloxegol Tablets, 25 mg and of a Naloxegol Solution Formulation, 25 mg, Compared to Whole Naloxegol Tablets, 25 mg, in Healthy Subjects
Brief Title: A Bioavailability Study With Alternate Methods of Administration of Naloxegol Tablets, and Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00035
Record Dates: First submitted 2015-04-29; First posted 2015-05-18 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Bioavailability; Healthy Subjects
Keywords: naloxegol tablet crushed; naloxegol oral solution; naloxegol whole tablet; relative bioavailability; Phase I; healthy subjects
MeSH Terms: interventions — naloxegol; Tablets; Excipients; Water; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatments A-D-B-C sequence (Experimental): Treatment A in Period 1, Treatment D in Period 2, Treatment B in Period 3 and Treatment C in Period 4
  Interventions: Drug: Naloxegol 25 mg tablet, crushed, suspended in water, given orally; Drug: Naloxegol 25mg tablet crushed, suspended in water, given via nasogastric tube; Drug: Naloxegol 25 mg (10 mL oral solution); Drug: Naloxegol 25 mg tablet, given orally
- Treatments B-A-C-D sequence (Experimental): Treatment B in Period 1, Treatment A in Period 2, Treatment C in Period 3 and Treatment D in Period 4
  Interventions: Drug: Naloxegol 25 mg tablet, crushed, suspended in water, given orally; Drug: Naloxegol 25mg tablet crushed, suspended in water, given via nasogastric tube; Drug: Naloxegol 25 mg (10 mL oral solution); Drug: Naloxegol 25 mg tablet, given orally
- Treatments C-B-D-A sequence (Experimental): Treatment C in Period 1, Treatment B in Period 2, Treatment D in Period 3 and Treatment A in Period 4
  Interventions: Drug: Naloxegol 25 mg tablet, crushed, suspended in water, given orally; Drug: Naloxegol 25mg tablet crushed, suspended in water, given via nasogastric tube; Drug: Naloxegol 25 mg (10 mL oral solution); Drug: Naloxegol 25 mg tablet, given orally
- Treatments D-C-A-B sequence (Experimental): Treatment D in Period 1, Treatment C in Period 2, Treatment A in Period 3 and Treatment B in Period 4
  Interventions: Drug: Naloxegol 25 mg tablet, crushed, suspended in water, given orally; Drug: Naloxegol 25mg tablet crushed, suspended in water, given via nasogastric tube; Drug: Naloxegol 25 mg (10 mL oral solution); Drug: Naloxegol 25 mg tablet, given orally

INTERVENTIONS:
Drug: Naloxegol 25 mg tablet, crushed, suspended in water, given orally — naloxegol 25 mg (1 tablet) crushed, suspended in water, given orally
  Other Names: Treatment A; (Test product)
Drug: Naloxegol 25mg tablet crushed, suspended in water, given via nasogastric tube — naloxegol 25 mg (1 tablet) crushed, suspended in water, given via nasogastric tube
  Other Names: Treatment B; (Test product)
Drug: Naloxegol 25 mg (10 mL oral solution) — naloxegol 25 mg (10 mL oral solution)
  Other Names: Treatment C; (Test product)
Drug: Naloxegol 25 mg tablet, given orally — naloxegol 25 mg (1 tablet) whole tablet, given orally
  Other Names: Treatment D; (Reference product)

SUMMARY:
This clinical study is an open-label, randomized, 4-period, 4-treatment, crossover, single-center, single-dose bioavailability study with alternate methods of administration of crushed naloxegol tablets, 25 mg and of a naloxegol solution formulation, 25 mg, compared to whole naloxegol tablets, 25 mg, in healthy subjects.

The main objective of this study is to determine the bioavailability of each of three alternative methods of naloxegol administration compared to whole naloxegol tablets given orally by assessment of the primary pharmacokinetic (PK) parameters of naloxegol

DETAILED DESCRIPTION:
This is an open-label, randomized, 4-period, 4-treatment, crossover, single-center, single-dose bioavailability study with alternate methods of administration of naloxegol: crushed and suspended in water and administered orally (Treatment A),crushed and suspended in water administered via nasogastric tube (Treatment B), solution administered orally (Treatment C) and tablet swallowed as a whole (Treatment D).

Alternative ways of administering a tablet may be useful to help patients who, for different reasons, have difficulties with swallowing a whole tablet. Administration of dispersed (crushed) tablets suspended in water is a common way of administering drugs to these patients. A useful method in patients whose condition prevents swallowing is administration of dispersed tablets through nasogastric tubes. Additionally a solution formulation may be an attractive option for some patients including the pediatric population. The main aim in this clinical study is to investigate whether the blood concentrations of naloxegol (pharmacokinetic) after each treatment A, B and C is comparable to that after treatment D. Additionally, the safety and tolerability shall be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the clinical unit, must not be lactating and must be of non childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  * Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy; but not tubal ligation.
* Have a body mass index (BMI) between 18.5 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Able to understand, read and speak the German language.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influence the results or the potential subject's ability to participate in the study.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

Drugs include known CYP3A4 and/or P-gp inhibitors and inducers, e.g., diltiazem, verapamil, and erythromycin

- Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.

For females, hormonal replacement therapy is not allowed.

* Subject with a relevant history of a suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 6 months (a level of 4 or 5), or who are at significant risk to commit suicide, as judged by the investigator using the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Applicable to subjects willing to participate in genetic research: Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL International GmbH, Berlin
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- [Background] Bui K, Birmingham B, Diva U, Berger B. An Open-Label, Randomized Bioavailability Study of Alternative Methods of Oral Administration of Naloxegol in Healthy Subjects. Clin Pharmacol Drug Dev. 2017 Jul;6(4):420-427. doi: 10.1002/cpdd.335. Epub 2017 Jan 27. PMID 28127938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL International, Early Phase Clinical Unit Berlin, Berlin, Germany.
Pre-assignment Details: Participants were randomized in 4 sequence Williams design for 4 periods and 4 treatments: 25 mg naloxegol tablet crushed and suspended in water taken orally(Treatment A), 25 mg naloxegol tablet crushed and suspended in water via nasogastric tube (Treatment B), 2.5 mg/mL oral solution (Treatment C) and 25 mg naloxegol tablet swallowed(Treatment D).
Groups:
- ADBC Sequence: Treatment A in Period 1, Treatment D in Period 2, Treatment B in Period 3 and Treatment C in Period 4.
- BACD Sequence: Treatment B in Period 1, Treatment A in Period 2, Treatment C in Period 3 and Treatment D in Period 4.
- CBDA Sequence: Treatment C in Period 1, Treatment B in Period 2, Treatment D in Period 3 and Treatment A in Period 4.
- DCAB Sequence: Treatment D in Period 1, Treatment C in Period 2, Treatment A in Period 3 and Treatment B in Period 4.
Period: Overall Study
Arm/Group | ADBC Sequence | BACD Sequence | CBDA Sequence | DCAB Sequence
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 9 | 11
Not Completed | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADBC Sequence | BACD Sequence | CBDA Sequence | DCAB Sequence | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 42 (11) | 45 (8) | 44 (8) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 3 | 11
  Male | 8 | 9 | 8 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-infinity).
Description: Area under plasma concentration-time curve from time zero extrapolated to infinity (AUC) is presented below. Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: Pre-dose (0 hours [within 30 minutes prior to administration of the investigational medicinal product (IMP)]) and post-dose at 0.25 (15 minutes), 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours in each treatment period.
Population: The Pharmacokinetic (PK) analysis set was a subset of those participants in the safety analysis set and included participants who had received at least 1 dose of study medication and had at least 1 post-dose plasma concentration measurement at a scheduled time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Treatment A: Participants received Naloxegol 25 mg oral tablet, crushed, suspended in water.
- Treatment B: Participants received Naloxegol 25 mg crushed, suspended in water, given via nasogastric tube.
- Treatment C: Participants received Naloxegol 25 mg of 10 mL oral solution.
- Treatment D: Participants received Naloxegol 25 mg whole tablet orally.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
h*ng/mL | 191 (54.2) | 192 (48.0) | 179 (54.0) | 191 (47.2)
Statistical Analysis 1: Comparison: Treatment A vs Treatment D; Test type: Superiority or Other; ANOVA; The results are based on ANOVA of log transformed PK parameters with sequence, period, treatment, and subject nested within sequence as fixed effects; Ratio# = 98.89, 90% CI 2-sided [92.40 to 105.84]
Statistical Analysis 2: Comparison: Treatment B vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 100.04, 90% CI 2-sided [93.17 to 107.43]
Statistical Analysis 3: Comparison: Treatment C vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 94.37, 90% CI 2-sided [88.70 to 100.40]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC 0-t).
Description: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration is presented below. Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: Pre-dose (0 hours [within 30 minutes prior to IMP administration]) and post-dose at 0.25 (15 minutes), 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours in each treatment period.
Population: The PK analysis set was a subset of those participants in the safety analysis set and included participants who had received at least 1 dose of study medication and had at least 1 post-dose plasma concentration measurement at a scheduled time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
h*ng/mL | 188 (54.4) | 190 (47.8) | 178 (53.7) | 188 (47.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 98.79, 90% CI 2-sided [92.24 to 105.80]
Statistical Analysis 2: Comparison: Treatment B vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 100.44, 90% CI 2-sided [93.65 to 107.72]
Statistical Analysis 3: Comparison: Treatment C vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 94.83, 90% CI 2-sided [89.20 to 100.82]

3. Primary Outcome: Observed Maximum Plasma Concentration (Cmax).
Description: Observed maximum plasma concentration (Cmax) is presented below. Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
ng/mL | 39.2 (44.1) | 40.1 (45.1) | 40.2 (45.7) | 39.7 (51.8)
Statistical Analysis 1: Comparison: Treatment A vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 97.05, 90% CI 2-sided [88.09 to 106.92]
Statistical Analysis 2: Comparison: Treatment B vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 100.56, 90% CI 2-sided [91.80 to 110.16]
Statistical Analysis 3: Comparison: Treatment C vs Treatment D; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio# = 102.5, 90% CI 2-sided [93.13 to 111.82]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax).
Description: This was one of the PK parameters to determine the time to reach maximum plasma concentration (tmax). Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 42 | 41 | 43
h | 0.75 [0.23 to 5.00] | 1.50 [0.25 to 5.02] | 0.50 [0.25 to 5.00] | 1.00 [0.23 to 5.03]

5. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz).
Description: This was one of the PK parameters to determine λz of a t½λz. Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
h | 9.92 (3.92) [0.23 to 5.00] | 8.78 (4.22) [0.25 to 5.02] | 9.28 (3.40) [0.25 to 5.00] | 9.22 (3.13) [0.23 to 5.03]

6. Secondary Outcome: Mean Dissolution Time (MDT).
Description: This was one of the PK parameters to determine MDT (whole tablet only) (calculated as MRT Treatment D [Reference] - MRT Treatment C [Test]). Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: as for outcome 2
Population: The PK analysis set was a subset of those participants in the safety analysis set and included participants who had received at least 1 dose of study medication and had at least 1 post-dose plasma concentration measurement at a scheduled time point. There were zero participants analyzed in Treatment A, B and C, hence data was not determined.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment D
Number analyzed (Participants) | 26
h | 1.29 (0.951) [0.23 to 5.03]

7. Secondary Outcome: Mean Residence Time (MRT).
Description: This was one of the PK parameters to determine MRT. Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
h | 6.94 (2.00) [0.23 to 5.00] | 6.54 (1.92) [0.25 to 5.02] | 6.21 (1.42) [0.25 to 5.00] | 6.72 (1.68) [0.23 to 5.03]

8. Secondary Outcome: Apparent Total Body Clearance After Extravascular Administration Estimated as Dose Divided by AUC (CL/F).
Description: This was one of the PK parameters to determine the apparent total body clearance after extravascular administration estimated as dose divided by AUC. Blood was collected pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose to determine naloxegol plasma concentrations.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
L/h | 131 (54.2) [0.23 to 5.00] | 130 (48.0) [0.25 to 5.02] | 140 (54.0) [0.25 to 5.00] | 131 (47.2) [0.23 to 5.03]

9. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F).
Description: This was one of the PK parameters to determine the apparent volume of distribution during the terminal phase after extravascular administration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 41 | 40 | 43
L | 1738 (55.3) [0.23 to 5.00] | 1513 (55.4) [0.25 to 5.02] | 1731 (58.5) [0.25 to 5.00] | 1640 (54.7) [0.23 to 5.03]

10. Secondary Outcome: Percentage of Participants With Adverse Events (AE).
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.The term AE is used generally to include any AE whether serious or non-serious. An serious AE (SAE) is an AE that fulfills one or more of the following criteria: results in death, is immediately life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; is a congenital abnormality or birth defect; is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: For up to 9 weeks (starting with screening).
Population: The safety analysis set included all participants who had received at least one dose of Naloxegol and for whom any safety post-dose data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
percentage of participants | 9.5 | 7.0 | 11.6 | 18.6

11. Secondary Outcome: Mean Change From Baseline for Vital Signs of Supine Systolic and Diastolic Blood Pressure.
Description: The following variables were collected after the participants had rested in the supine position for at least 5 minutes: Systolic Blood Pressure (SBP) and Diastolic BP. The measurement of vital signs for SBP and DBP are presented in the below outcome table.
Time Frame: Day 2 (24h post-dose), Day 3 (48h post-dose) and Day 4 (72h post-dose).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
mmHg
  Day 2/24h Post-dose (SBP) (N= 42, 43, 43, 43) | -2 (9) | -4 (11) | -1 (8) | 0 (8)
  Day 3/48h Post-dose (SBP) (N= 42, 43, 43, 42) | 4 (9) | -2 (10) | 2 (8) | 2 (8)
  Day 4/72h Post-dose (SBP) (N= 9, 11, 11, 12) | 7 (9) | 0 (9) | 1 (11) | 7 (13)
  Day 2/24h Post-dose (DBP) (N= 42, 43, 43, 43) | -2 (6) | -4 (7) | -1 (5) | 0 (6)
  Day 3/48h Post-dose (DBP) (N= 42, 43, 43, 42) | 0 (6) | -2 (7) | 0 (6) | 1 (5)
  Day 4/72h Post-dose (DBP) (N= 9, 11, 11, 12) | 5 (7) | 0 (6) | 4 (3) | 4 (6)

12. Secondary Outcome: Mean Change From Baseline for Vital Signs in Supine Pulse Rate.
Description: Pulse rate: the measurement of vital signs for pulse rate is presented in the below outcome table.
Time Frame: Day 2 (24h post-dose), Day 3 (48h post-dose) and Day 4 (72h post-dose).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
beats per minute (bpm)
  Day 2/24h Post-dose (N= 42, 43, 43, 43) | 1 (5) | 0 (6) | 1 (6) | 2 (6)
  Day 3/48h Post-dose (N= 42, 43, 43, 42) | 5 (6) | 4 (7) | 5 (8) | 5 (6)
  Day 4/72h Post-dose (N= 9, 11, 11, 12) | 8 (9) | 4 (9) | 8 (5) | 12 (5)

13. Secondary Outcome: Participants With Significant Findings in Physical Examination.
Description: A complete physical examination included an assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, mouth and throat), lymph nodes, thyroid, musculoskeletal and neurological systems. Physical examination was performed to check for any significant abnormality in participants.
Time Frame: A full physical examination at screening and the final follow-up visit (maximum 9 weeks apart). Abbreviated physical examination on admission (on Day -1 of each treatment period) and at 48-hours post-dose to each treatment period (for up to 4 weeks).
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Participants With Significant Findings in Columbia-Suicide Severity Rating Scale (C-SSRS).
Description: The C-SSRS is a unique, simple and short method of assessing both behavior and ideation that tracks all suicidal events, and provided a summary of suicidality. It assesses the lethality of attempts and other features of ideation (frequency, duration, controllability, reasons for ideation and deterrents), all of which are significantly predictive of completed suicide. The C-SSRS was performed to determine the presence of suicidality.
Time Frame: At Baseline and Days 1-4 of each treatment period.
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Participants With Significant Findings in 12-Lead Electrocardiography (ECG).
Description: A 12-lead ECG was obtained after the participant rested in supine position for at least 10 minutes. The study physician was to judge the overall interpretation as normal or abnormal. If abnormal, it was decided as to whether or not the abnormality was clinically significant and the reason for the abnormality was recorded.
Time Frame: At screening, first admission to the clinical unit (Visit 2, Day -1), 1.25 hours after each dose (Visits 2-5, Day 1), as well as at the final follow-up visit (up to 9 weeks).
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Participants With Significant Findings in Hematology, Clinical Chemistry and Urinalysis.
Description: Participants were assessed through each laboratory variables for any significant abnormalities. Hematology assessments included white blood cell count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin and others. Clinical chemistry assessment included testing levels of sodium, potassium, urea, creatinine, albumin, calcium, glucose (fasting) and others. Urinalysis assessment included glucose, protein, blood and microscopy (if positive for blood or protein).
Time Frame: At screening and at the final follow-up visit (maximum 9 weeks apart); in addition, for the first and third treatment period at pre-dose.
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 42 | 43 | 43 | 43
participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Taste Test Assessment.
Description: A standardized questionnaire was provided to participants and were asked to complete the questionnaire for the liquid formulations tested, i.e., Naloxegol crushed tablet, oral (Treatment A) and Naloxegol oral solution (Treatment C), without assistance or influence from site personnel. For each formulation, the questionnaire was identical and required the participant's opinion. Sweet, salty, sour, bitter, metallic, hot/spicy were rated on a scale of 0 to 10, where 0 means not at all and 10 means extreme. The overall rating of the taste was rated on a scale of 0 to 10, where 0 means "I dislike it extremely much" and 10 means "I like it extremely much". The smell of the medicine was based on a scale of 0 to 10, where 0 means extremely bad and 10 means extremely nice. The question on whether the participants would consider ever taking the medicine again was based on a scale of 0 to 10, where 0 means "Never - under no circumstances" and 10 means "Yes, definitely".
Time Frame: Within 1 hour after dosing (Treatments A and C only).
Population: as for outcome 10
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 42 | 43
units on a scale
  Sweet | 0.0 (0.0) [0 to 2] | 7.0 [1 to 10]
  Salty | 0.0 [0 to 7] | 0.0 [0 to 4]
  Sour | 0.0 [0 to 5] | 0.0 [0 to 6]
  Bitter | 3.0 [0 to 8] | 0.0 [0 to 5]
  Metallic | 1.0 [0 to 7] | 0.0 [0 to 4]
  Hot/Spicy | 0.0 [0 to 1] | 0.0 [0 to 2]
  How would you rate the taste of this medicine? | 4.0 [0 to 8] | 7.0 [1 to 10]
  If the medicine smells, how does it smell? | 4.0 [3 to 5] | 7.0 [5 to 9]
  Would you consider taking this medicine again? | 8.0 [0 to 10] | 9.0 [1 to 10]

ADVERSE EVENTS:
Time Frame: SAEs were reported from the signing of the informed consent and AEs were recorded from randomization until the final follow-up/ early-termination visit.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 4/42 | 3/43 | 5/43 | 8/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=42) | Treatment B (N=43) | Treatment C (N=43) | Treatment D (N=43)
Headache (Nervous system disorders) | 1 | 1 | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.